CLINICAL TRIAL: NCT04181619
Title: Influence of Coffeeberry Extract on Soccer Specific Skill Performance After Rest, During Simulated Soccer Match Play, and Following Fatiguing Exercise in Academy Football Players
Brief Title: Influence of Coffeeberry Ingestion on Soccer Skill Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1904
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Skill Performance; Soccer Performance; Coffeeberry Effects
Keywords: coffeeberry; caffeine; polyphenols; chlorogenic acid; exercise; soccer; skill; performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffeeberry beverage (Experimental): 300 mg Coffeeberry extract in 300 ml beverage
  Interventions: Dietary Supplement: Coffeeberry beverage
- Color and flavor matched beverage (Placebo Comparator): 0 mg Coffeeberry extract in 300 ml flavor and color-matched beverage
  Interventions: Other: Comparator beverage

INTERVENTIONS:
Dietary Supplement: Coffeeberry beverage — One exposure of 300 mg coffeeberry extract in a 300 ml flavored still beverage prior to exercise session
  Arms: Coffeeberry beverage
Other: Comparator beverage — One 300 ml still beverage, color and flavor matched to experimental beverage prior to exercise session
  Arms: Color and flavor matched beverage

SUMMARY:
The study of soccer skill performance has 3 objectives. Objective 1 is to compare effects of coffeeberry (300mg) and placebo ingestion on dribbling speed and precision and passing and shooting speed and accuracy compared to placebo. 30 subjects will be assessed before dosing, after a 1 hr resting absorption period, and after simulated soccer match play. Of these 30, 20 subjects will proceed to Objective 2 (45 minutes of intense simulated soccer match play) and Objective 3 (repeated sprint activity continued until volitional fatigue).

ELIGIBILITY:
Inclusion Criteria:

* Provide valid informed consent prior to any study procedure
* Male soccer players age 16 to 28 years
* 5-year soccer playing experience
* 1-year regularly soccer training
* Free of injuries
* Willing to avoid alcohol in the 48-h period prior to main trials.
* Willing to avoid caffeine, caffeinated and decaffeinated products, apples, and, berries/cherries for 24-h prior to main trials
* Willing to record food intake over the 48-h period prior to the first trial and replicate for second trial
* Willing to abstain from strenuous physical activity for 24-h before all visits

Exclusion Criteria:

* Smoking
* Cardiovascular diseases
* Diabetes or other metabolic disease
* Presence of injuries
* Major illnesses or surgery in prior 90 days
* Participation in another clinical trial in the past month

Ages: 16 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Dribbling speed | During 3.5 hours post consumption
  m/sec, increase would be better. Simulated match in an indoor gym with pre-set targets.
Dribbling precision | During 3.5 hours post consumption
  Meters, more accuracy would be better. Simulated match in an indoor gym against pre-set targets.
Passing accuracy | During 3.5 hours post consumption
  1-10 scale, higher score would be better. Simulated match in an indoor gym against pre-set targets.
Passing speed by Time | During 3.5 hours post consumption
  km/h, increased would be better. Simulated match in an indoor gym against pre-set targets.
Shooting accuracy | During 3.5 hours post consumption
  More shots on target would be better. Simulated match in an indoor gym against pre-set targets.
Shooting speed | During 3.5 hours post consumption
  Milliseconds, faster would be better. Simulated match in an indoor gym against pre-set targets.

SECONDARY OUTCOMES:
Sprint speed | During 3.5 hours post consumption
  m/sec, increase would be better. In indoor gym with marked course.
High-intensity endurance running capacity | During 3.5 hours post consumption
  Run time to volitional fatigue in min, increase would be better. In indoor gym with marked course.

OTHER OUTCOMES:
Blood analyte concentration: Capillary glucose | During 3.5 hours post consumption
  (mmol/L), more regulated would be better
Blood analyte concentration: Capillary lactate | During 3.5 hours post consumption
  (mmol/L), lower (delayed rise) would be better
Blood analyte concentration: Serum chlorogenic acid | During 3.5 hours post consumption
  (mmol/L), n.a. for placebo, introduced to evaluate primary outcomes
Blood analyte concentration: Serum caffeine | During 3.5 hours post consumption
  (ug/mL), n.a. for placebo, Introduced to evaluate primary outcomes
Rate of Perceived Exertion (RPE) | During 3.5 hours post consumption
  By Borg scale, rated 6-20, lower values would be better
Activation/Deactivation (feelings and mood) | During 3.5 hours post consumption
  Checklist of feelings using a 4 point scale from definitely do to definitely don't feel, more relaxed and better mood would be better
Mental energy | During 3.5 hours post consumption
  By Visual Analog Scale (VAS) vertical marking on 100 mm horizontal line, higher energy would be better
Physical energy | During 3.5 hours post consumption
  By Visual Analog Scale (VAS) vertical marking on 100 mm horizontal line, higher energy would be better
Heart rate | During 3.5 hours post consumption
  By electronic reading, lower would be better
Gut comfort | During 3.5 hours post consumption
  By Visual Analog Scale (VAS) vertical marking on 100 mm horizontal scale, no or less nausa, fullness or bloating would be better
Hydration status | During 3.5 hours post consumption
  Urine osmolality in mOsm/kg, comparing pre- vs. post-exercise concentration

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Galloway, PhD, Principal Investigator — U. Stirling
Locations (1):
- University of Stirling, Health Science and Sport, Stirling, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No